CLINICAL TRIAL: NCT01841762
Title: A Multi-center, Open-label, Single-arm, Phase 3b Study of Macitentan in Patients With Pulmonary Arterial Hypertension to Psychometrically Validate the PAH-SYMPACT Instrument
Brief Title: Clinical Study of Macitentan in Patients With Pulmonary Arterial Hypertension to Psychometrically Validate the PAH-SYMPACT Instrument
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-055-401
Record Dates: First submitted 2013-03-27; First posted 2013-04-29 (Estimated); Results first posted 2018-10-31 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH-SYMPACT; Pulmonary Arterial Hypertension; psychometric instrument
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Macitentan (Experimental): Macitentan tablet, dose of 10 mg, once daily
  Interventions: Drug: Macitentan

INTERVENTIONS:
Drug: Macitentan — Macitentan tablet, dose of 10 mg, once daily
  Other Names: Macitentan / ACT-064992

SUMMARY:
SYMPHONY is prospective, multi-center, open-label, single-arm, Phase 3b psychometric validation study of the PAH-SYMPACT, a new quality of life questionnaire for patients with pulmonary arterial hypertension. Patients will be in the study for 5 1/2 months, 4 months of which they will receive macitentan, 10 mg, once daily.

The primary objectives are to demonstrate the final content validity of the PAH SYMPACT instrument, to demonstrate the psychometric characteristics of reliability and construct validity of the PAH-SYMPACT instrument, and to demonstrate the ability of the PAH SYMPACT instrument to detect change. The secondary objective is to assess the safety of macitentan in patients with pulmonary arterial hypertension. The exploratory objective is to explore the effects of macitentan on PAH symptoms and their impact (as measured by the PAH-SYMPACT) in patients with pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to initiation of any study mandated procedure
2. Patients with symptomatic PAH in World Health Organization (WHO) Functional Class (FC) II to IV
3. Patients with PAH belonging to one of the following subgroups of the Dana Point Clinical Classification Group 1:

   1. Idiopathic, or
   2. Heritable, or
   3. Drug or toxin induced, or
   4. Associated with one of the following:

   i. Connective tissue disease ii. Congenital heart disease with simple systemic-to-pulmonary shunt at least one year after surgical repair iii. HIV infection
4. Documented hemodynamic diagnosis of PAH by right heart catheterization - performed at any time prior to Screening showing:

   1. Resting mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg and
   2. Resting pulmonary vascular resistance (PVR) > 240 dyn•s•cm-5 and
   3. Pulmonary capillary wedge pressure (PCWP) or left ventricular end diastolic pressure (LVEDP) ≤ 15 mmHg
5. 6-minute walk distance (6MWD) ≥ 150 m at Screening
6. Able to fluently speak and read English
7. For patients on phosphodiesterase type-5 inhibitors (PDE5i), inhaled prostacyclin analogues, or calcium channel blockers, stable doses for at least 3 months prior to Visit 2
8. For patients on oral diuretics, stable doses for at least 4 weeks prior to Visit 2
9. Men or women aged 18 or older

   1. A woman is considered to be of childbearing potential unless she:

      * Has not yet entered puberty, or
      * Does not have a uterus, or
      * Has gone through menopause (has not had a period for at least 12 months for natural reasons, or who has had their ovaries removed)
   2. A women of childbearing potential is eligible only if she meets both criteria below:

      * Has a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline and agree to perform monthly urine pregnancy tests, and
      * Agrees to use two methods of contraception (one method for patients with a progesterone implant or an intrauterine device or tubal sterilization) from the Screening Visit 1 until one month after study drug discontinuation

Exclusion Criteria:

1. Moderate to severe obstructive lung disease: forced expiratory volume in one second (FEV1) / forced vital capacity < 70% and FEV1 < 65% of predicted value after bronchodilator administration
2. Moderate to severe restrictive lung disease: total lung capacity < 60% of predicted value
3. Hemoglobin < 75% of the lower limit of the normal range at screening
4. Serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3 times the upper limit of normal (ULN) at screening
5. Estimated creatinine clearance < 30 mL/min at screening
6. Systolic blood pressure (SBP) < 90 mmHg at screening
7. Body weight < 40 kg at screening
8. Known concomitant life-threatening diseases with a life expectancy of < 12 months
9. Any condition that prevents compliance with the protocol or adherence to therapy
10. Treatment with endothelin receptor antagonists (ERAs) within 3 months prior to Visit 2, or scheduled to receive any of these compounds, other than macitentan, during the trial
11. Treatment with intravenous or subcutaneous prostacyclin or prostacyclin analogs within 3 months prior to Visit 2, or scheduled to receive any of these compounds during the trial
12. Treatment with riociguat within 3 months prior to Visit 2, or scheduled to receive riociguat during the trial
13. Treatment with strong cytochrome P450 (CYP) 3A4 inducers or inhibitors within 4 weeks prior to Visit 2
14. Recently started (< 8 weeks prior to Visit 2) or planned cardio-pulmonary rehabilitation program based on exercise
15. Females who are lactating or pregnant (positive Screening or Baseline pregnancy test) or plan to become pregnant during the study
16. Known hypersensitivity to macitentan or its excipients or drugs of the same class
17. Treatment with another investigational drug within 3 months prior to Visit 2
18. Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results such as drug or alcohol dependence or psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2015-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Romero, PharmD, PhD, Study Chair — Actelion Pharmaceuticals US, Inc; Gary Palmer, MD, MBA, Study Chair — Actelion Pharmaceuticals US, Inc.
Locations (81):
- United States (81):
  - Cardiovascular Associates of the Southeast, LLC, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pulmonary Associates, PA, Phoenix, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - UCSF Fresno, Fresno, California
  - UCSD Medical Center, Pulmonary Department, La Jolla, California
  - VAGLAHS, VA Greater LA Healthcare System, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - Los Angeles Biomedical Research Institute, Torrance, California
  - University of Colorado, Aurora, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Bay Area Cardiology Associates, P.A., Brandon, Florida
  - University of Florida Academic Health Center, Gainesville, Florida
  - University of Florida College of Medicine, Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Georgia Regents University, Augusta, Georgia
  - Georgia Clinical Research, Austell, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical, Chicago, Illinois
  - Advocate Health and Hospitals Corporation, Oakbrook Terrace, Illinois
  - Chest Infectious Diseases and Critical Care Associates, PC, Des Moines, Iowa
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Iowa City Heart Center, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Veritas Clinical Specialties, Topeka, Kansas
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Beaumont Hospital, Troy, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Midwest Pulmonary Consultants, Kansas City, Missouri
  - Ferrell-Duncan Clinic, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Clinic Pulmonology, St Louis, Missouri
  - Clayton Sleep Institute, St Louis, Missouri
  - Nebraska Pulmonary Specialties, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Pulmonary and Critical Care Associates, Union, New Jersey
  - Buffalo General Medical Center, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - North Shore-LIJ/Advance Lung Disease Clinic, New Hyde Park, New York
  - Beth Israel Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, Weiler Division, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Novant Health Pulmonary and Critical Care, Matthews, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - UC Health/University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Davis Heart & Lung Research Institute, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - The Oregon Clinic, Portland, Oregon
  - CDA for Oregon Pulmonary Associate, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University, Division on Pulmonary and Critical Care, Philadelphia, Pennsylvania
  - Temple Lung Center, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Berks Schuylkill Respiratory Specialists, Ltd., Wyomissing, Pennsylvania
  - Wellspan Lung, Sleep and Critical Care, York, Pennsylvania
  - Sioux Falls Cardiovascular, PC, Sioux Falls, South Dakota
  - Baylor Research Institute (BRI), Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Inova Heart and Vascular Institue / Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Pulmonary & Sleep Research, Spokane, Washington
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Chin KM, Gomberg-Maitland M, Channick RN, Cuttica MJ, Fischer A, Frantz RP, Hunsche E, Kleinman L, McConnell JW, McLaughlin VV, Miller CE, Zamanian RT, Zastrow MS, Badesch DB. Psychometric Validation of the Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT) Questionnaire: Results of the SYMPHONY Trial. Chest. 2018 Oct;154(4):848-861. doi: 10.1016/j.chest.2018.04.027. Epub 2018 Apr 26. PMID 29705220

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy-nine sites recruited subjects to reach a total of 284 total enrolled, with 335 subjects entered screening. Institution-based and community clinic sites, with pulmonary arterial hypertension expertise, were included in the study. The first subject, first visit occurred on 25 APR 2013 and last subject, last visit occurred on 05 OCT 2015
Pre-assignment Details: Screen failures total 51 subjects. Six subjects were removed from the full analysis set of 284 due to exclusion. The per protocol set includes 278 subjects total (97.9% of enrollment), utilized for all validation and exploratory ePRO analyses. The safety set, encompassing all enrolled subjects receiving study treatment, includes 284 subjects.
Period: Screening Period
Arm/Group | Macitentan
Started | 335
Completed | 284
Not Completed | 51
Not completed — Other, 2 PAH-SYMPACT cycles not complete | 51
Period: Treatment Period
Arm/Group | Macitentan
Started | 284
Completed | 252
Not Completed | 32
Not completed — Adverse Event | 16
Not completed — Death | 1
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 2
Not completed — Other, including non-compliance | 5
Period: Post-Treatment Safety Follow-Up Period
Arm/Group | Macitentan
Started | 284
Completed | 269
Not Completed | 15
Not completed — Death | 1
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 6
Not completed — Other, administrative error | 1

BASELINE CHARACTERISTICS:
Population: The number of subjects who dosed on macitentan in the trial was 284.
Arm/Group | Macitentan
Number analyzed (Participants) | 284
Age, Categorical [Count of Participants; unit: Participants] — Age of patients reported.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 167
    >=65 years | 117
Age, Continuous [Mean (Inter-Quartile Range); unit: Years] — Full Analysis Set of 284 patients. Population: Each respective row population complies with overall number of patients.
  Years | 59.7 [52.0 to 69.0]
Sex: Female, Male [Count of Participants; unit: Participants] — A total of 284 participants analyzed.
  Participants
    Female | 223
    Male | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — A total of 284 participants analyzed.
  Participants
    Hispanic or Latino | 27
    Not Hispanic or Latino | 257
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — A total of 284 participants analyzed.
  Participants
    American Indian or Alaska Native | 2
    Asian | 8
    Native Hawaiian or Other Pacific Islander | 1
    Black or African American | 35
    White | 228
    More than one race | 10
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Development and Refinement of the Patient-reported Outcome Measure of Symptoms and Their Impact in PAH (the PAH-SYMPACT)
Description: Content validity of the PAH-SYMPACT was assessed using item performance, exploratory and confirmatory factor analysis. The final item content and domain structure of PAH-SYMPACT was determined based on these analyses from the Steering Committee (expert clinicians) and findings from the qualitative research done with patients previously.
Time Frame: From Screening Visit (Day -14) to End of Treatment (EOT) Visit (Visit 4, Week 16)
Population: Per Protocol Set (PPS) comprised all patients included in the Full Analysis Set (FAS) who had no major protocol violations.
Measure: Number; unit: Items
Arm/Group | Macitentan
Number analyzed (Participants) | 278
Items
  Item number in symptoms part of baseline | 16
  Item number in symptoms part at Week 16 | 11
  Item number in impacts part at baseline | 25
  Item number in impacts part at Week 16 | 11

2. Primary Outcome: Validation of the Patient-reported Outcome Measure of Symptoms and Their Impact in PAH (the PAH-SYMPACT), With Reliability Assessed Via Test-retest Reliability.
Description: The reliability of the PAH-SYMPACT is assessed by test-retest reliability. Intra-class correlation coefficients (ICCs) assess test-retest reliability for the symptom and impact part scores as well as domains. ICCs equal to or greater than 0.70 are considered to demonstrate good test-retest reliability for total and domain scores.
Time Frame: From ePRO period 1 (Days -14 to -8) to ePRO period 2 (Days -7 to -1) in screening period.
Population: Per Protocol Set of 278 patients.
Measure: Number; unit: Intra-class correlation coefficient
Arm/Group | Macitentan
Number analyzed (Participants) | 278
Intra-class correlation coefficient
  ICCs of Cardiopulmonary Symptoms domain | 0.94
  ICCs of Cardiovascular Symptoms domain | 0.93
  ICCs of Physical Impacts domain | 0.91
  ICCs of Cognitive/Emotional Impacts domain | 0.84

3. Primary Outcome: Validation of the Patient-reported Outcome Measure of Symptoms and Their Impact in PAH (the PAH-SYMPACT), Assessing Internal Consistency Reliability.
Description: The reliability of the PAH-SYMPACT is assessed by internal consistency reliability. This was determined using Cronbach's alpha-a value on an internal level scale from 0 to 1.0 with higher scores indicating a more-reliable (precise) instrument.
Time Frame: From ePRO period 1 (Days -14 to -8) to ePRO period 2 (Days -7 to -1) in screening period.
Population: Per protocol set of 278.
Measure: Number; unit: Ratio of variance
Arm/Group | Macitentan
Number analyzed (Participants) | 278
Ratio of variance
  Cronbach's Alpha for Cardiopulmonary Symptoms | 0.81
  Cronbach's Alpha for Cardiovascular Symptoms | 0.88
  Cronbach's Alpha for Physical Impacts Domain | 0.92
  Cronbach's Alpha for Cognitive/Emotional Impacts | 0.87

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events, Serious Adverse Events, and Adverse Events Resulting in Patient Study Drug Discontinuation Between Time Periods, BL to End of Study Visit (EoS, Week 16+30 Days for Follow-up Safety Visits)
Description: Safety events are reported and documented as defined in study protocol.
Time Frame: From Day 1 (Baseline Visit) to End of Study visit (EoS).
Population: Safety set of 284 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan
Number analyzed (Participants) | 284
Participants
  Participants with AEs | 228
  Participants with severe intensity AEs | 36
  Participants with SAEs | 49
  Participants prematurely discontinued study drug | 17

5. Other Pre Specified Outcome: Assessment of the Sensitivity to Detect Change in the Symptoms and Impacts Domain Scores of the PAH-SYMPACT From Baseline to Week 16.
Description: Sensitivity to change is an aspect of construct validity and represents the instrument's ability to detect underlying change. Sensitivity to change was examined to compare the difference in mean score in each domain of the PAH-SYMPACT. The symptoms and impacts domains consisted of 11 items each reported on a 7-point Likert Scale (from 0=no symptom/with no difficulty at all/not at all to 6=very severe symptoms/very much/extremely/not able at all). An average symptoms domain score is determined based on the daily scores of the containing items. An average impacts domain score is determined based on the items in the domain.
Time Frame: From Screening period (Days -7 to -1) to Week 16 (7-day period prior to Week 16 visit).
Population: Per Protocol Set of 278 subjects.
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Macitentan
Number analyzed (Participants) | 278
Score on a scale
  Cardiopulmonary Symptoms domain score at baseline | 1.0 [0.5 to 1.3]
  Cardiopulmonary Symptoms domain score at Week 8 | 0.8 [0.4 to 1.2]
  Cardiopulmonary Symptoms domain score at Week 16 | 0.7 [0.4 to 1.2]
  Cardiovascular Symptoms domain score at baseline | 0.4 [0.1 to 0.7]
  Cardiovascular Symptoms domain score at Week 8 | 0.2 [0.0 to 0.5]
  Cardiovascular Symptoms domain score at Week 16 | 0.2 [0.0 to 0.5]
  Physical Impacts domain score at baseline | 1.3 [0.6 to 2.0]
  Physical Impacts domain score at Week 8 | 1.0 [0.4 to 1.7]
  Physical Impacts domain score at Week 16 | 0.9 [0.4 to 1.6]
  Cogn./Emotional Impacts domain score at baseline | 0.8 [0.3 to 1.5]
  Cogn./Emotional Impacts domain score at Week 8 | 0.8 [0.3 to 1.3]
  Cogn./Emotional Impacts domain score at Week 16 | 0.5 [0.5 to 1.3]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from study drug initiation until Day 30 after study drug discontinuation.
Description: Study sites were instructed to document any adverse change from the patient's baseline condition, i.e., any unfavorable and unintended sign, including an abnormal laboratory finding, symptom, or disease that occurs during the course of the study, whether or not considered related to the study drug. Counts and percentages of subjects who experienced adverse events were tabulated by system organ class and preferred term within each system organ class, as well as by individual preferred term.
Arm/Group | Macitentan
All-Cause Mortality (participants affected / at risk) | 1/284
Serious Adverse Events (participants affected / at risk) | 49/284
Other Adverse Events (participants affected / at risk) | 228/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan (N=284)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Chest Pain (General disorders) | 4
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 3
Cardiac Failure (Cardiac disorders) | 3
Cardiac Failure Congestive (Cardiac disorders) | 3
Fluid Overload (General disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Renal Failure Acute (Renal and urinary disorders) | 3
Small Intestinal Obstruction (Gastrointestinal disorders) | 3
Acute Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 2
Diverticulitis (Gastrointestinal disorders) | 2
Hypoglycaemia (Blood and lymphatic system disorders) | 2
Transfusion (Surgical and medical procedures) | 2
Vertigo (Nervous system disorders) | 2
Angina Unstable (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Atrial Flutter (Cardiac disorders) | 1
Bladder Transitional Cell Carcinoma (Renal and urinary disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan (N=284)
Oedema peripheral (Blood and lymphatic system disorders) | 50
Headache (Nervous system disorders) | 36
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34
Cough (Respiratory, thoracic and mediastinal disorders) | 26
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 23
Fatigue (General disorders) | 22
Dizziness (Ear and labyrinth disorders) | 19
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 19
Nausea (General disorders) | 17
Anaemia (Blood and lymphatic system disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Actelion for review at least 30 days prior to submission for publication or presentation. Upon review, Actelion may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights. Neither the institution nor the investigator should permit publication during such a review period.